CLINICAL TRIAL: NCT04782973
Title: A Novel Disease Management Platform Delivered Via Smartphone Application for the Management of Patients With Heart Failure: Pilot Study
Brief Title: Disease Management Platform for Heart Failure (DMP-HF)
Acronym: DMP-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Pradeep Natarajan, Director, Preventive Cardiology, Assistant Professor of Medicine, Harvard Medical School, Associate Member of the Broad Institute of Harvard and MIT, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P004027
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — isofenphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group - AMAZE™ Disease Management Platform (Other): Eligible patients 21+ years with a diagnosis of HF admitted to MGH cardiology services. The intervention group is exposed to the AMAZE™ app for 60 days. Participants will interact with a nurse for a 7-day discharge follow-up call, a medication reconciliation, assess understanding of heart meds, assess patients' HF symptoms, provide tailored guidance, set goals related to medication adherence, exercise, diet, and other health behaviors. The nurse will coordinate with cardiology teams to streamline med refills, cardiology appointments, and cardiac rehabilitation referrals. The nurse and patient will connect via telephone and in-app messaging, to address patients' concerns and state of health.
  Interventions: Other: AMAZE (TM) Disease Management Platform

INTERVENTIONS:
Other: AMAZE (TM) Disease Management Platform — Providing patients with smartphone app that will integrate with provider facing dashboard within electronic medical record.

SUMMARY:
AMAZE™ is a disease management platform (DMP) designed to educate patients about heart failure, help engage them in healthy behaviors and assist them in taking their medications as prescribed. This study will assess whether the AMAZE™ smartphone-based application ("app") can help heart failure patients take better care of themselves after discharge from an inpatient heart failure admission at Massachusetts General Hospital (MGH).

The primary objective is to demonstrate feasibility and perceived value of the AMAZE™ platform in clinical practice. The study will also explore whether the use of the AMAZE™ platform for 60 days post-discharge leads to a reduction in hospital readmission, emergency department, urgent care and unexpected ambulatory care visits. The impact of the AMAZE™ platform on participant reported quality of life outcomes and perception of overall medical care will also be examined.

DETAILED DESCRIPTION:
Heart failure (HF) management and readmissions remain at the top of the list of complex topics in cardiovascular medicine in the United States. Current system-wide programs to curb HF-related hospital readmissions have shown inconsistent results. However, outpatient transitional care supportive programs have been linked to improved HF-related outcomes, including reduced hospital readmissions, in small studies. Small studies also indicate that remote transfer of non-invasive data through telemonitoring (e.g., blood pressure and weight) and structured telephone support may reduce hospital readmissions in a cost-effective manner. The present pandemic has placed significant strains on the link between clinicians and patients highlighting the need for rapid innovation for virtual care.

This study involves the AMAZE™ DMP, developed by AstraZeneca, to provide a unified experience for the management of HF patients throughout their patient care journey. The platform will integrate multiple systems, including a smartphone-based application where patients can enter daily mood, symptoms, weight measures, and vital signs such as blood pressure (BP) and medication adherence. This input will feed directly to a clinician facing dashboard embedded within the electronic medical record that will allow the clinical care team to access real-time views of patients' states both in and out of clinic.

Patients will be identified via an automated electronic medical record (EMR)-based, computer-based algorithm and eligibility will be manually verified. Participants will be enrolled in the study following an inpatient HF admission at Massachusetts General Hospital (MGH).

Clinical providers and study staff will be able to view and monitor the subjects' AMAZE™ smartphone application entries within the electronic medical record via the AMAZE™ provider dashboard. The AMAZE™ secure messaging function will be used for study and clinical communications between the patient, study staff and clinical care team to facilitate outpatient HF management. The AMAZE™ smartphone application (app) will indirectly assess the patient's quality of life (Kansas City Cardiomyopathy Questionnaire - KCCQ), as well as patient satisfaction with the app (mHealth App Usability Questionnaire - MAUQ). For clinicians, the MAUQ will measure provider satisfaction with the AMAZE™ dashboard.

Baseline demographics and study outcomes will be assessed via direct patient survey by study staff at pre-specified time points (enrollment, 30-days post enrollment, 60-days post enrollment). Outcomes will include medication changes, hospitalizations, emergency department presentations, urgent care visits, primary care or cardiology office visits and cardiac rehabilitation enrollment. Medical history, including labs, procedures, and diagnoses will be collected from the electronic medical record and recorded in REDCap. The AMAZE™ app will track medication adherence, daily symptom(s) log, blood pressure, weight, heart rate and activity when entered by participants into a daily log. Participants will be asked and encouraged to enter information into the smartphone-based app daily by study staff.

The primary goal of the present proposal will be to generate evidence on the feasibility and perceived value of the AMAZE™ platform implemented in clinical practice. The outcomes will be measured using conversion rate (study enrollment rate among total number of eligible patients) and utilization rate (percentage of days participants engaged with the AMAZE™ app during the 60-day study period). This study is a first necessary step before testing efficacy in a large multi-center study.

ELIGIBILITY:
Inclusion Criteria:

Adults (>21 years) admitted to MGH Cardiology services (Ellison 10 and 11) with a primary diagnosis of heart failure [HFrEF(<40%), HFmEF(40-49%) HFpEF(≥50%)] (or to BWH Cardiology services for BWH EHR-based controls)

Has a smartphone or iPad and is willing to enter health metrics into DMP App and email willing to use for the study

Access to the internet

Established or with plan to establish primary cardiologist at MGH (or at BWH for BWH EHR-based controls)

Discharged home or to self-care (with or without home services)

Exclusion Criteria:

Moderate or severe cognitive impairment

Non-English-speaking

Palliative management only (comfort measures)

Does not own a smartphone or iPad (not considered for EHR-based controls)

Incarcerated

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Natarajan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Over the 6-months 2,071 patients were screened. Of these, 409 were considered eligible for the study. Staff approached 167 patients. A total of 70 patients consented to participate. A total of 51 out of 70 enrolled patients completed the study. Common reasons patients declined were study felt like it might be too much work (n=51), did not feel comfortable using smartphone (n=17), requested time to consider, but could not be contacted (n=10). Declined to provide a reason (n=10)
Groups:
- Intervention Group - AMAZE™ Disease Management Platform: The intervention group was exposed to the AMAZE™ app for 60 days, following discharge from the hospital. Patients were consented once eligibility was confirmed. During the 60-day period, patients were expected to complete daily logs of wellbeing, heart failure symptoms, physical activity levels, medication adherence, weight, blood pressure, and heart rate. Patients were prompted to complete the KCCQ and MAUQ within the app at set timepoints.
  AMAZE™ contained curated links to articles about heart failure causes, diagnosis, and management which patients could access at will. Patients received a 7-day discharge follow-up call from the nurse navigator. The nurse completed a medication reconciliation and assessed and expanded the patients' understanding of their heart medications. The nurse asked questions about the patients' heart failure symptoms and provided guidance for symptom monitoring and management, discussed lifestyle modifications and assisted in setting goals related to medication adherence, exercise, diet, and other health behaviors. The nurse coordinated with the patients' clinical care team, streamlining med refills, cardiology appointments, and cardiac rehab referrals. Subsequent correspondences between the nurse and patient took place by telephone and in-app messaging for the duration of the study period. The nurse navigator addressed patients' concerns, questions, and state of health as represented by data entered by the patients into the app.
Period: Overall Study
Arm/Group | Intervention Group - AMAZE™ Disease Management Platform
Started | 70
Completed | 51
Not Completed | 19
Not completed — Withdrawal by Subject | 5
Not completed — Protocol Violation | 6
Not completed — No Longer Eligible Post-Consent | 8

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group - AMAZE™ Disease Management Platform
Number analyzed (Participants) | 51
Age, Customized [Mean (Standard Deviation); unit: years]
  Age Mean | 65.9 (12.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 36
  Female | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46
  Black | 3
  Asian | 0
  Other | 2
  Unknown | 0
Clinical conditions and co-morbidities [Number; unit: participants]
  Hypertension | 45
  Coronary artery disease | 39
  Hyperlipidemia | 36
  Atrial fibrillation | 29
  Anemia | 26
  Depression | 25
  Chronic kidney disease | 19
  Chronic lung disease | 18
  Obstructive sleep apnea | 18
  Diabetes | 16
  Cancer | 11
  Cerebrovascular disease | 10
  Thyroid disorder | 10
  Peripheral artery disease event | 9
  Abdominal aortic aneurysm | 3
  Familial hypercholesterolemia | 3
  Cirrhosis | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Implementation
Description: Feasibility of implementing the AMAZE™ platform is assessed in terms of the number of patients who completed the study.
Time Frame: 6 months
Population: English-speaking patients aged 21 years and older who carried a chart diagnosis of heart failure with established or planned longitudinal cardiovascular care at MGH
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: Patients admitted to MGH Cardiology floors considered eligible following manual chart review of their electronic medical records.
- Approached Patients: Eligible patients who were approached for recruitment to the study
- Enrolled Patients: Patients who consented to participating in the study
Arm/Group | Eligible Patients | Approached Patients | Enrolled Patients
Number analyzed (Participants) | 409 | 167 | 70
Participants | 51 | 51 | 51

2. Primary Outcome: Perceived Value of Disease Management Platform
Description: Perceived value was measured using the participants' scoring of the platform's features in the mHealth App Usability Questionnaire (MAUQ). The questionnaire has 21 questions, with scores were based on a scale of 1 (disagree) to 7 (agree).
Time Frame: 60 days
Population: Of 51 completed participants, 21(41.2%) completed the 60-day MAUQ.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group - AMAZE™ Disease Management Platform
Number analyzed (Participants) | 21
score on a scale
  The app was easy to use | 6 [6 to 7]
  It was easy for me to learn to use the app | 7 [6 to 7]
  I like the interface of the app | 6 [4.5 to 7]
  The information in the app was well organized, so I could easily find the information I needed | 6 [5 to 6]
  I feel comfortable using this app in social settings | 6 [6 to 7]
  The amount of time involved in using this app has been fitting for me | 6 [6 to 7]
  I would use this app again | 6 [6 to 7]
  Overall, I am satisfied with this app | 6 [5.5 to 6]
  Whenever I made a mistake using the app, I could recover easily and quickly | 6 [5 to 6.5]
  This mHealth app provides an acceptable way to receive healthcare services | 6 [5 to 6]
  The app adequately acknowledged and provided information to let me know the progress of my action | 6 [4 to 6]
  The navigation was consistent when moving between screens | 6 [6 to 7]
  The interface of the app allowed me to use all the functions offered by the app | 6 [5 to 6]
  This app has all the functions and capabilities I expected it to have | 6 [5 to 6]
  The app would be useful for my health and wellbeing | 6 [5 to 7]
  The app improved my access to healthcare services | 6 [5 to 7]
  The app helped me manage my health effectively | 6 [5 to 6]
  The app made it convenient for me to communicate with my healthcare provider | 6 [4.5 to 6]
  Using the app, I had many more opportunities to interact with my healthcare provider | 6 [4 to 6]
  I felt confident that any information I sent to my provider using the app would be received | 6 [6 to 6.5]
  I felt comfortable communicating with my healthcare provider using the app | 6 [4.5 to 7]

3. Secondary Outcome: Disease Management Platform Engagement
Description: Participants' engagement with the platform was measured in terms of daily logs completed and number of messages sent to the nurse navigator.
Time Frame: 60 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention Group - AMAZE™ Disease Management Platform
Number analyzed (Participants) | 51
days
  Number of days participants engaged with the platform during the first 30 days of the study period | 22 [11 to 28]
  Number of days participants engaged with the platform over the 60-day study period | 44 [14 to 53]

4. Secondary Outcome: Health Status Change With Use of Disease Management Platform
Description: Health status was ascertained based on participants' responses to the Kansas City Cardiomyopathy Questionnaire-12 (KCCQ), which assesses heart failure symptoms and impact on quality of life. The questionnaire was administered at baseline, 30 days after enrolling in the study, and 60 days after enrolling in the study. Change in health status was measured by the difference in scores between the first and last KCCQ completed (baseline and 60 days after). KCCQ scores range from 0 (very poor health) to 100 (excellent health). An increase in score indicates improvement in health status and a decrease indicates worsening health status. The measure we use here reports the change in KCCQ scores from a 15-point decrease to a 15-point increase from baseline in increments of 5 points.
Time Frame: 60 days
Population: Of the 51 participants who completed the study, 29 participants completed at least two surveys of the baseline and 30- and 60-day KCCQs.
Measure: Number; unit: participants
Arm/Group | Intervention Group - AMAZE™ Disease Management Platform
Number analyzed (Participants) | 29
participants
  Number of participants whose score decreased by at least 15 points | 2
  Number of participants whose score decreased by at least 10 points | 2
  Number of participants whose score decreased by at least 5 points | 5
  Number of participants whose score did not change | 6
  Number of participants whose score increased by at least 5 points | 18
  Number of participants whose score increased by at least 10 points | 9
  Number of participants whose score increased by at least 15 points | 9

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events over the 60-day study period.
Groups:
- Intervention Group - AMAZE™ Disease Management Platform: Over the six-month recruitment period (03/2021-09/2021) there are no adverse events to report for the 70 participants enrolled.
Arm/Group | Intervention Group - AMAZE™ Disease Management Platform
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT04782973/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT04782973/ICF_001.pdf